CLINICAL TRIAL: NCT04818034
Title: The Effect of Sodium-glucose Cotransporter (SGLT) 2 Inhibitors on Cystine Stone Formation: A Preliminary Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGLT2
Record Dates: First submitted 2021-03-17; First posted 2021-03-26 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Cystinuria
MeSH Terms: conditions — Cystinuria | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 10 mg Dapagliflozin taken orally once daily for 4 weeks (Experimental): 10 mg of the study drug Dapagliflozin taken orally once daily for 4 weeks
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin is to lower blood sugar levels in adults with type 2 diabetes.
  Other Names: FARXIGA

SUMMARY:
Cystinuria is an inherited autosomal recessive disorder of the kidney that is the result of an inability to reabsorb cystine from the urine. Supersaturation of cystine in the urine produces crystals that precipitate and form stones in the kidney, which can be a cause of obstruction, infection, and chronic kidney disease. Cystine stones constitute a major health challenge for affected individuals with cystinuria because of the frequent recurrence of painful symptoms and the current absence of effective, patient-accepting treatment.

A mainstay of therapy is breaking or preventing the cystine bond on the molecular level such that cystine (which is formed from the joining of two cysteine amino acids and their corresponding sulfur atoms) cannot precipitate in the urine. It is hypothesized that a glucose molecule may be able to do this if introduced into the urine. SGLT-2 inhibitors are a class of drug that are FDA approved to treat diabetes mellitus (DM) and heart failure by inhibiting an enzyme in the kidney that allows for reabsorption of glucose from the urine. This effectively increases the concentration of glucose in the urine. Our hypothesis suggests that administration of this drug to patients with cystine will introduce sufficient glucose into the urine to prevent the formation of cystine stones. To date, there has been no published data on the effectiveness of this therapy for this indication, although the dosage and administration would be identical to that already approved by the FDA for the treatment of DM and heart failure.

DETAILED DESCRIPTION:
This is a single center, proof of concept prospective cohort trial designed to assess the effect of daily oral administration of dapagliflozin on cystine formation in freshly voided urine. Five subjects are planned, each with previously diagnosed cystinuria and without current treatment except with potassium citrate medication.

Total duration of subject participation with be up to four weeks. Total duration of the study is expected to be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* males and females age 18 or older
* documented cystinuria on prior 24-hour urine collection and/or stone analysis
* history of previous cystine kidney stones
* able and willing to provide consent

Exclusion Criteria:

* prior diagnosis of diabetes mellitus (type I or type II)
* current SGLT-2 inhibitor administration at the time of screening
* SGLT-2 inhibitor administration within the last year prior to screening
* vulnerable populations including incarceration status
* anticipation of pregnancy during the study duration
* unable to give informed consent
* non-English primary language
* pregnancy, lactation, or child- bearing age without birth control devices
* serious illness likely to cause death within the next 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Stoller, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study team will identify the patients being treated for cystinuria within the study team's clinic. The study team will inform these patients of the study and provide them with the study details to allow further discussion and to answer any questions the patients might have.
Pre-assignment Details: There is only one arm for this study. Any patient willing to participate in this study will be in that arm and will be given the study drug Dapagliflozin.
Groups:
- Study Drug: The study drug Dapagliflozin
Period: Overall Study
Arm/Group | Study Drug
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Drug
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: 24hr Urine Measurements of the Effect of SGLT-2 Inhibitor Therapy on Cystine Production in Urine in Patients With Cystinuria
Description: The primary efficacy endpoint will be assessed by comparing previous 24hr urine cystine concentration data collected prior to study participation and 24hr urine concentration data collected after being on the study drug, specifically examining the content of cystine in the urine but not exclusively.
Time Frame: 1 month
Population: The analysis was specifically looking at cystine production in urine but other products were analyzed as well as shown in the table.
Measure: Mean (Standard Deviation); unit: 24hr urine cystine concentration (mg)
Arm/Group | Study Drug
Number analyzed (Participants) | 10
24hr urine cystine concentration (mg) | 999.3 (1.1)
Statistical Analysis 1: Comparison: Study Drug; Test type: Other — paired t-test; p = 0.965, paired t-test; paired t-test = 0.965, Standard Deviation 37

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow-up, 4 weeks.
Arm/Group | Study Drug
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Our study has several important limitations. First, this was a retrospective study with a limited follow up duration on SGLT2 inhibitors. Second, treating the stone event rate as its own control may introduce healthcare utilization bias as interfacing with the medical system could have led to improved dietary habits which had a major impact on stone event rates. Third, patients with cystinuria are known to develop symptomatic calculi in clusters for unknown reasons. The sample size is small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT04818034/Prot_SAP_000.pdf